CLINICAL TRIAL: NCT01014195
Title: Risk of Psychopathology and Neurocognitive Impairment in Leukemia Survivors
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: NEULS; R01MH085849 (NIH)
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Neurocognitive Impairment; Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Neurocognitive function; ADHD; brain imaging; genetic polymorphisms; Psychopathology and neurocognitive Impairment in Leukemia Survivors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Survivors of pediatric leukemia treated on Total Therapy Protocol XV (TOTXV) at St. Jude Children's Research Hospital (SJCRH), who are ≥ 8 years of age and ≥ 5 years from diagnosis.
  Intervention: Neurocognitive and behavioral evaluation
  Interventions: Other: Neurocognitive and behavioral evaluation

INTERVENTIONS:
Other: Neurocognitive and behavioral evaluation — The primary neurocognitive outcome will be performance on measures of cognitive flexibility and cognitive fluency. Functional behavior will be evaluated via the child or adult version of the Behavior Rating Inventory of Executive Function, using parent respondent for each version. The presence of ADHD and common comorbid conditions (i.e. depression, anxiety) will be determined with structured diagnostic interviews. Quality of life will be re-assessed with the PedQL.

SUMMARY:
1. This study will evaluate the association between changes in basic cognitive and behavioral functioning by the end of chemotherapy treatment, and the later development of higher order executive functions in pediatric acute lymphoblastic leukemia (ALL).
2. The association between acute treatment-related changes in brain integrity and subsequent brain maturation in long-term survivors of pediatric ALL will be evaluated.
3. The association between patterns of behavioral and executive dysfunction and brain maturation in long-term survivors of pediatric ALL will be examined.
4. The association between genetic polymorphisms in key enzyme pathways and higher order brain development in long-term survivors of pediatric ALL will be explored.
5. The associations between biologic and behavioral indices of fatigue/sleep and higher order brain development in long-term survivors of pediatric ALL will be explored.

DETAILED DESCRIPTION:
Survival rates for pediatric acute lymphoblastic leukemia (ALL) now exceed 80%. With this growing population of long-term survivors comes recognition that a considerable proportion experience one or more significant late effects. For children undergoing central nervous system (CNS) treatment, common late effects include neurocognitive impairment and neurobehavioral problems. Although these problems first manifest as subtle difficulties with attention and processing speed, they can evolve into deficits in higher order brain functions that significantly impact functional skills in a subset of long-term survivors. There currently is no method to accurately identify patients at greatest risk for these long-term behavioral and neurocognitive problems. Through this proposal, this study plans to utilize existing data collected during acute treatment to identify predictors of long-term neurocognitive and brain maturation outcomes. The study also proposes to collect data on attention-deficit/hyperactivity disorder (ADHD) and associated comorbidities, higher order executive functions, and structural and functional brain imaging in survivors who are at least 8 years of age and greater than 5 years from diagnosis.

All patients will undergo a single neurocognitive evaluation focused on assessment of higher order executive functions. Patients will be evaluated during their regularly scheduled annual follow-up visit, when health-related monitoring will also occur. Parents of participants will be asked to complete questionnaires designed to assess the family environment and the impact of cancer diagnosis on family functioning and parent stress.

Brain Imaging: To better demonstrate untoward treatment effects upon cortical brain development, quantitative MR imaging of myelin integrity using diffusion tensor imaging (DTI) and cortical thickness assessment using high resolution volumetric imaging will be utilized. All patients will also be evaluated using functional MRI (fMRI) procedures during resting state and participation in attention and working memory tasks. fMRI and DTI data will be de-identified then analyzed at MD Anderson Cancer Center in Houston, Texas.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled on SJCRH TOTXV ALL protocol
* ≥ 5 years post diagnosis of ALL
* ≥ 8.0 years of age at time of follow-up evaluation

Exclusion Criteria:

* History of cranial or total-body radiation therapy
* History of bone marrow transplant
* History of relapse
* History of head injury, neurological condition unrelated to ALL treatment, or diagnosis of a genetic disorder associated with neurocognitive impairment (e.g. Down Syndrome)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children originally enrolled and treated on the SJCRH TOTXV protocol. The study has reviewed TOTXV patient database and has identified 343 patients (189 males and 154 females) who will meet the inclusion criteria (assuming no additional deaths or relapse).
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2010-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Neurocognitive assessment of attention, processing speed, and executive functions. | Once, at least 5 years post ALL diagnosis and 2 years off treatment

SECONDARY OUTCOMES:
Quantitative magnetic resonance imaging (MRI) and DTI and functional magnetic resonance imaging (fMRI) of brain structure and function. | Once, at least 5 years post ALL diagnosis and 2 years off treatment
Family and parental stress as reported by primary caregiver. | Once, at least 5 years post ALL diagnosis and 2 years off treatment
Associations between genetic polymorphisms in key enzyme pathways and higher order brain development in long-term survivors of pediatric ALL. | Once, at least 5 years post ALL diagnosis and 2 years off treatment
Associations between fatigue and neurocognitive performance and between sleep problems and neurocognitive performance. | Once, at least 5 years post ALL diagnosis and 2 years off treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Krull, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Cheung YT, Sabin ND, Reddick WE, Bhojwani D, Liu W, Brinkman TM, Glass JO, Hwang SN, Srivastava D, Pui CH, Robison LL, Hudson MM, Krull KR. Leukoencephalopathy and long-term neurobehavioural, neurocognitive, and brain imaging outcomes in survivors of childhood acute lymphoblastic leukaemia treated with chemotherapy: a longitudinal analysis. Lancet Haematol. 2016 Oct;3(10):e456-e466. doi: 10.1016/S2352-3026(16)30110-7. Epub 2016 Sep 14. PMID 27658980
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols